CLINICAL TRIAL: NCT05324735
Title: Pentoxifylline for Treatment of Resistant Major Depression: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Pentoxifylline for Treatment of Resistant Major Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Talar A. Merza Mohammad, Associate Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMU PE-EC 24112021/391
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Resistant Major Depression
Keywords: Bipolar Depression; Pentoxifylline; Resistant Major Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline (tablet): 400 mg twice a day for 12 weeks
  Interventions: Drug: Pentoxifylline
- Control group (Placebo Comparator): Placebo (tablet): twice a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — All participants will receive pentoxifylline 400 mg (orally ingested) twice a day for 12 weeks.
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — All participants will receive placebo (orally ingested) twice a day for 12 weeks.
  Other Names: Sugar Pills
  Arms: Control group

SUMMARY:
A growing body of evidence has highlighted the role of inflammation and phosphodiesterases (PDE)-related pathways in the pathogenesis of neuropsychiatric illnesses such as depression/mood disorders. Herein, we aimed to evaluate the therapeutic benefits of pentoxifylline (PTX) in the treatment of therapy-resistant depression (TRD) in adult patients with bipolar depression.

DETAILED DESCRIPTION:
Depression, which affects an estimated 300 million people worldwide, is the main cause of mental health-related illness burden. Depression keeps people from attaining their full potential, depletes human capital, and is linked to suicide and other forms of mortality. Despite the fact that depressive disorders have a better prognosis than primary psychotic illnesses like schizophrenia, 20%-40% of patients treated with antidepressants do not respond to their initial treatment regimens, and up to 15% do not respond to multiple antidepressant regimens and modalities, such as electroconvulsive shock (ECT) therapy. Since the treatment resistance has been shown to increase the likelihood of full symptomatic recurrence, worsen the treatment course and quality of life; therefore, there is a critical need for innovative treatment techniques for patients who have failed to respond to traditional treatments. Inflammation is one factor that has gotten a lot of attention lately as an etiologic mechanism of treatment-resistant depression (TRD). Increased levels of (pro) inflammatory markers such as tumor necrosis factor-alpha (TNF-α), interleukin (IL)-1, and IL-6 are reported in a considerable percentage of patients with major depressive disorders with or without other comorbidities, including bipolar depression and TRD patients. Also, clinical factors connected to antidepressant response are linked to the reduction of inflammatory cytokines.

Moreover, cytokine antagonists, such as the chimeric anti-TNF-alpha antibody infliximab, has shown antidepressant efficacy. Hence, given the elevated levels of inflammatory activity in TRD patients, new treatments with anti-inflammatory effect might be an effective approach to treat these patients. Pentoxifylline (PTX) is a methylated xanthine derivative that has been used to treat peripheral vascular disease for more than two decades. PTX has anti-inflammatory and phosphodiesterase (PDE) inhibitory effects that enables it to inhibit PDEs competitively. Subsequently, it can increase cAMP levels, activate protein kinase A (PKA), inhibit ILs and TNF-α production, and reduce inflammation. Therefore, PTX-decreased inflammatory activity, may give rapid symptomatic alleviation for medically healthy individuals with TRD depression.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, voluntary informed consent prior to study enrollment.
* Male or female between the ages of 18 to 65.
* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-IV) criteria for bipolar I or II, currently experiencing a major depressive episode. A Mini-International Neuropsychiatric Interview (MINI) conducted by physician was used to confirm the diagnosis.
* Meets the criteria for treatment resistant depression (TRD) defined by failure to respond to of at least two treatment trials (antidepressant regimen or electroconvulsive therapy) during the current depressive episode.
* Prior to taking part in the trial, all patients were requested to be antidepressant free for 4 weeks or to be on a fixed psychotropic therapeutic regimen for at least 4 weeks.

Exclusion Criteria:

* Current psychotic symptoms or perceptual problems.
* The presence of a contraindication to PTX, such as a drug allergy or xanthine derivative allergy.
* Patients with substance dependence or abuse.
* Patients with concurrent active medical condition (congestive heart failure, abnormal electrocardiogram, malignancy, schizophrenia, neurological disease).
* Patients with inflammatory disorders and/or auto-immune conditions (rheumatoid arthritis, inflammatory bowel disease, multiple sclerosis, lupus)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale-17 (HAM-D-17) Scores | 12 weeks
  The HAM-D-17 is a 17-item scale that asks participants to rate the severity of their depression symptoms. Scoring is based on the 17-item scale. The total score ranges from 0 to 52, with higher numbers demonstrating more severe symptoms. Normal scores range from 0 to 7, mild depression ranges from 8 to 16, moderate depression ranges from 17 to 23, and scores of 24 and greater indicate severe depression. Remission is defined as HAM-D-17 total score ≤ 7 (primary outcome).

SECONDARY OUTCOMES:
Response Rate | 12 weeks
  The number of patients with a ≥ 50% drop in the Hamilton Depression Rating Scale-17 (HAM-D-17) total score.
Remission Rate | 12 weeks
  The number of patients reaching depression remission. Remission is defined as Hamilton Depression Rating Scale-17 (HAM-D-17) total score ≤ 7.
Serum level of CRP | 12 weeks
  Peripheral blood samples will be collected to assess changes in the serum levels of C- reactive protein (mg/dl).
Serum level of TNF-α | 12 weeks
  Peripheral blood samples will be collected to assess changes in the serum levels of tumor necrosis factor alpha (pg/ml).
Serum level of IL-6 | 12 weeks
  Peripheral blood samples will be collected to assess changes in the serum levels of Interleukin-6 (pg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Talar A Merzamohammad, Pharm. D, Principal Investigator — Hawler Medical University, College of Pharmacy, Department of Pharmacology and Toxicology
Locations (1):
- Hawler Psychiatric Hospital and Private Clinic, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No